CLINICAL TRIAL: NCT00834665
Title: Phase I/II Combination Immunotherapy After ASCT for Advanced Myeloma to Study HTERT Vaccination Followed by Adoptive Transfer of Vaccine-Primed Autologous T Cells
Brief Title: Phase I/II Clinical Trial Combining hTERT Tumor Vaccine & Autologous T Cells in Patients With Advanced Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Maryland, College Park (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 13406 / GCC610
Record Dates: First submitted 2008-01-03; First posted 2009-02-03 (Estimated); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- hTERT/GM-CSF+PCV, T cell infusion (Experimental): ARM A = hTERT/GM-CSF+PCV, T cell infusion
  Interventions: Biological: hTERT vaccine, GM-CSF, PCV, T cell infusion
- GM-CSF+PCV, T cell infusion,GM-CSF+PVC (Experimental): ARM B GM-CSF+PCV, T cell infusion,GM-CSF+PVC
  Interventions: Biological: GM-CSF, PCV, T cell infusion

INTERVENTIONS:
Biological: hTERT vaccine, GM-CSF, PCV, T cell infusion — hTERT vaccine (multi-peptide vaccine), Granulocyte Macrophage-Colony Stimulating Factor (GM-CSF), Prevnar-Pneumococcal Conjugate vaccine (PCV), T cell infusion
  Arms: hTERT/GM-CSF+PCV, T cell infusion
Biological: GM-CSF, PCV, T cell infusion — Granulocyte Macrophage-Colony Stimulating Factor (GM-CSF), Prevnar-Pneumococcal Conjugate vaccine (PCV), T cell infusion
  Arms: GM-CSF+PCV, T cell infusion,GM-CSF+PVC

SUMMARY:
The purpose of this study is:

1. To evaluate the safety of activated T cell infusions and immunization with hTERT multi-peptide vaccine in the post-transplant setting and whether the combination can delay hematopoietic recovery or induce other autoimmune events.
2. To determine whether the strategy of infusing vaccine-primed T-cells early after transplant in conjunction with post-transplant boosters leads to the induction of cellular immune responses to hTERT.

DETAILED DESCRIPTION:
This protocol proposes to combine two different investigational products to test the hypothesis that autologous T cell therapy can augment the potency of a putative tumor vaccine post- stem cell transplant, and lead to a myeloma-directed T-cell mediated "graft vs. myeloma" effect in patients with advance myeloma. The hope is that this combination therapy approach will result in a more rapid recovery of acquired immunity and consequently increased cure rates and better clinical outcomes. The two investigational products to be evaluated in this Phase I/II study include:

1. hTERT Vaccine (the putative tumor vaccine)- a multi-peptide vaccine consisting of 3 peptides against the catalytic subunit of telomerase (hTERT D988Y, I540, and R572Y), 1 survivin peptide (Sur1M2- an antiapoptotic protein), and 1 CMV (cytopeptide (N495).
2. T cell therapy- T-cells isolated from the patient and activated/expanded ex vivo by antiCD3/28 beads.

This is a two-site study at the University of Pennsylvania and University of Maryland to recruit a total of fifty-six study patients. The key eligibility criteria are patients who have systemic or multifocal myeloma requiring autologous stem cell transplantation. After enrollment, patients will be divided into two arms (A and B) according to their HLA A2 status (A = HLA A2 +, B = HLA A2-). Patients in ARM A will be initially immunized with the hTERT vaccine along with a pneumococcal conjugate vaccine (PCV); patients in ARM B will be initially immunized and given boosters of PCV only. All patients will undergo T-cell harvest, stem cell mobilization and collection, high-dose chemotherapy, autologous stem cell transplant (ASCT), and an infusion of expanded T cells at day 2 after ASCT. Patients in ARM A will then receive three hTERT/PCV vaccine boosters at day 14, 42, and 90 after ASCT.

ELIGIBILITY:
Each subject must meet ALL of the following criteria during screening to be enrolled in the study:

1. Written informed consent must be obtained from all patients before entry into the study
2. Patients must have a diagnosis of myeloma
3. Patients must meet one of the following criteria:

   * Myeloma has relapsed, progressed, or failed to respond after at least one prior course of therapy.
   * Myeloma has responded partially to initial therapy but neither a complete nor a near-complete response has developed after at least 3 cycles or months of initial therapy.
   * Myeloma has high-risk features
4. Patients must have measurable disease on study entry.
5. Patients must be between ages 18-80 (inclusive).
6. Patients should have adequate vital organ function.
7. ECOG performance status 0-2
8. Women of child-bearing potential (WOCBP) and their spouses or partners must be willing to use adequate contraception for the duration of the active treatment phase of the study and for at least 4 months after the last dose of chemotherapy. In addition, contraceptive measures must be continued as long as the patient remains on maintenance thalidomide in accordance with the STEPS program.

Key Exclusion Criteria

Subjects who meet ANY of the following criteria cannot be enrolled in the study:

1. Pregnant or nursing females
2. HIV, HTLV-1/2 seropositivity
3. Known history of myelodysplasia
4. Known history of chronic active hepatitis or liver cirrhosis (if suspected by laboratory studies, should be confirmed by liver biopsy).
5. Active Hepatitis B
6. Prior autotransplant or allogeneic transplant
7. More than 4 distinct, prior courses of therapy for myeloma
8. History of severe autoimmune disease requiring steroids or other immunosuppressive treatments.
9. Active immune-mediated diseases including: connective tissue diseases, uveitis, sarcoidosis, inflammatory bowel disease, multiple sclerosis.
10. Evidence or history of other significant cardiac, hepatic, renal, ophthalmologic, psychiatric, or gastrointestinal disease which might increase the risks of participating in the study
11. Active bacterial, viral or fungal infections.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2006-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Primary toxicity endpoint | 2 yrs
  Incidence of delayed hematopoietic recovery and the incidence of Grade 3 or greater autoimmune events

CONTACTS AND LOCATIONS:
Overall Officials: Carl H June, MD, Study Chair — University of Pennsylvania
Locations (2):
- United States (2):
  - Greenbaum Cancer Center, Baltimore, Maryland
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rapoport AP, Aqui NA, Stadtmauer EA, Vogl DT, Fang HB, Cai L, Janofsky S, Chew A, Storek J, Akpek G, Badros A, Yanovich S, Tan MT, Veloso E, Pasetti MF, Cross A, Philip S, Murphy H, Bhagat R, Zheng Z, Milliron T, Cotte J, Cannon A, Levine BL, Vonderheide RH, June CH. Combination immunotherapy using adoptive T-cell transfer and tumor antigen vaccination on the basis of hTERT and survivin after ASCT for myeloma. Blood. 2011 Jan 20;117(3):788-97. doi: 10.1182/blood-2010-08-299396. Epub 2010 Oct 28. PMID 21030558